CLINICAL TRIAL: NCT03313713
Title: Randomised Placebo-Controlled Clinical Trial to Assess the Medium-term Effect of 3 g/Day of a Beta-glucan on Lipid Profile, Glycemia and Intestinal Health, in Moderately Hypercholesterolemic Subjects
Brief Title: Beta-glucan Effects on Lipid Profile, Glycemia and inTestinal Health (BELT)
Acronym: BELT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Chief Internal Medicine Unit, University of Bologna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BELT_2016
Record Dates: First submitted 2017-10-08; First posted 2017-10-18 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — beta-Glucans

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-glucans (Active Comparator): Beta-glucans, 3 g per day, per 8 weeks, at breakfast
  Interventions: Dietary Supplement: Beta-glucans
- Placebo (Placebo Comparator): Placebo, 3 g per day, per 8 weeks, at breakfast
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-glucans — Placebo consumption at breakfast (3 g per day)
  Arms: Beta-glucans
Dietary Supplement: Placebo — Placebo consumption at breakfast (3 g per day)
  Arms: Placebo

SUMMARY:
This will be a randomized, placebo-controlled, clinical trial carried out on moderately hypercholesterolemic subjects who will consume 3 g per day of beta-glucans, in order to evaluate the effects on lipid profile, glycemia and intestinal function

DETAILED DESCRIPTION:
In order to assess the mid term effects of beta-glucans on lipid profile, glycemia and intestinal function, moderately hypercholesterolemic subjects will be involved in a cross-over study and supplemented for 8 weeks with 3 g/day of beta-glucans or placebo. The two intervention periods will be spaced by a 4 week washout period

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol between 200 and 240 mg/dL and/or LDL cholesterol between 130 and 190 mg/dL
* Triglycerides lower than 200 mg/dL
* Cardiovascular risk at 10 years lower than 10%
* Informed consent

Exclusion Criteria:

* Secondary prevention for cardiovascular diseases
* TG > 400 mg/dL, HDL-C < 35 mg/dL
* BMI higher than 30
* Assumption of lipid lowering drug or supplement with fibre or probiotics during the last 2 months
* Alcohol abuse
* Food allergy
* Alterations in thyroid, liver, or kidney functions, muscle diseases
* Diabetes, irritable bowel syndrome or chronic disturbed gut function

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
12 hour fasting lipid profile change from the baseline to the end of the intervention period | At the screening visit (4 weeks before the randomization one), at the randomization visit (week 0), after 4 and 8 weeks of treatment in both intervention periods (up to 24 weeks overall)
12 hour fasting glycemia change from the baseline to the end of the intervention period | At the screening visit (4 weeks before the randomization one), at the randomization visit (week 0), after 4 and 8 weeks of treatment in both intervention periods (up to 24 weeks overall)

SECONDARY OUTCOMES:
Intestinal function from the baseline to the end of the intervention period | At the screening visit (4 weeks before the randomization one), at the randomization visit (week 0), after 4 and 8 weeks of treatment in both intervention periods (up to 24 weeks overall)
  Intestinal function will be assessed by the use of a scale questionnaire investigating the number of weekly bowel movements, stool consistency, ease of defecation, sensation of emptying after defecation, intensity of discomfort during the defecation, feeling of bloating.
Liver function markers (glutamic oxalacetic transaminase, alanine transaminase, glutamic-pyruvic transaminase, aspartate transaminase) change from the baseline to the end of the intervention period | At the screening visit (4 weeks before the randomization one), at the randomization visit (week 0), after 4 and 8 weeks of treatment in both intervention periods (up to 24 weeks overall)
Blood pressure change from the baseline to the end of the intervention period | At the screening visit (4 weeks before the randomization one), at the randomization visit (week 0), after 4 and 8 weeks of treatment in both intervention periods (up to 24 weeks overall)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Borghi, MD, Principal Investigator — S. Orsola-Malpighi University Hospital
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided